CLINICAL TRIAL: NCT06900088
Title: Efficacy and Safety of Selinexor Combined With Azacitidine as Maintenance Therapy in High-Risk Myeloid Neoplasms Patients Post-Transplantation: A Single-Center, Single-Arm, Explorato
Brief Title: Selinexor Combined With Azacitidine Therapy in High-Risk Myeloid Neoplasms Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024099
Record Dates: First submitted 2024-12-27; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-12

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- patients with high-risk myeloid neoplasms after transplantation (Experimental): maintenance therapy with Selinexor combined with Azacitidine
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — maintenance therapy with Selinexor combined with Azacitidine in patients with high-risk myeloid neoplasms after transplantation

SUMMARY:
Efficacy and Safety of Selinexor Combined with Azacitidine as Maintenance Therapy in High-Risk Myeloid Neoplasms Patients Post-Transplantation: A Single-Center, Single-Arm, Exploratory Study

DETAILED DESCRIPTION:
Treatment period: From the time of transplantation, after screening by inclusion and exclusion criteria, patients who meet the criteria are enrolled and given maintenance therapy with Selinexor in combination with azacitidine (Selinexor: 40 mg/weekly, administered on D1; azacitidine: 50 mg/m2*5d; every 28 days for a cycle of treatment, for at least one year of medication, or until progression of the disease, or until the development of intolerable toxicity, whichever comes first)

ELIGIBILITY:
Inclusion criteria:

with pre-transplant MRD-positive AML, i.e., patients who meet one of the following criteria:

1. Age≥ 16 years old; any gender;
2. High-risk MDS (IPSS-R or/and IPSS-M high-risk and above);
3. High relapse risk AML, including relapsed refractory AML and patients with pre-transplant MRD-positive AML, i.e., patients who meet one of the following criteria:

(1)Refractory AML is defined as meeting one of the following conditions

1. Primary cases that have failed to respond to 2 courses of standard regimen chemotherapy;
2. CR was followed by consolidation and intensive treatment with no recurrence within 12 months;
3. It recurred 12 months later, but conventional chemotherapy was ineffective;
4. 2 or more relapses;
5. Extramedullary leukemia persists. (2)Relapsed AML i.e., re-initialization of leukemic cells in the peripheral blood after complete remission (CR) or bone marrow primitive cells >0.050 (except for other reasons such as bone marrow reconstitution after consolidation chemotherapy) or extramedullary infiltration of leukemic cells.

(3)Positive pre-transplant MRD, i.e., one of the following conditions is met:

1. Proportion of abnormal myeloid cells >0.01% by pre-transplant flow assay;
2. Positive pre-transplantation molecular biology-related tests. (4)AML with poor prognosis (according to the Chinese Guidelines for the Diagnosis and Treatment of Adult Acute Myeloid Leukemia (Non-Acute Promyelocytic Leukemia) 2023 Edition) 4.Meets WHO diagnostic criteria for staging CMML; 5.MDS or CMML transforms AML.

Exclusion criteria:

Patients with any of the following are not eligible for enrollment in this study:

1. Patients who relapsed within 3 months of transplantation or during maintenance therapy, including hematologic, molecular genetic, cytogenetic relapses, and extramedullary relapses.
2. Known positive serology for HIV or active hepatitis B virus (HBV) and hepatitis C virus (HCV);
3. Requirements for mental illness or other conditions that preclude cooperation with study treatment and monitoring;
4. Patients who are pregnant or who are unable to use appropriate contraception during treatment;
5. Suspected hypersensitivity to the experimental drug or any of its excipients;
6. Active heart disease, defined as one or more of the following:

（1）History of uncontrolled or symptomatic angina; （2）Myocardial infarction less than 6 months from study entry; （3）History of tardive dyskinesia requiring medication or clinically significant symptoms; （4）Uncontrolled or symptomatic congestive heart failure (> NYHA class 2) （5）Ejection fraction is below the lower limit of the normal range. 7. Those deemed unsuitable for enrollment by the investigator.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence free survival rate (RFS) | 2 years
  the rate at which a patient has been on the drug for at least 1 year without morphological relapse or death of the subject from the transplantation date (whichever comes first)

SECONDARY OUTCOMES:
2-year non-relapse mortality rate (NRM) | 2 years
  incidence of death from causes other than AML relapse/progression from the date of transplantation to the date of the subject's death
2-year survival rate (OS) | 2 years
  the 2-year survival rate from transplantation to death from any causes
Median overall survival (OS) | 2 years
  The time from transplantation to death from any causes
Cumulative incidence of acute graft-versus-host disease (GVHD) | 2 years
  Cumulative incidence of grade II-IV acute GVHD at 6 months after enrollment. Acute GVHD will be graded based on the diagnostic and severity scores used by the Blood and Bone Marrow Transplantation Clinical Trial Network (BMTCTN).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, China., Tianjin, China

IPD SHARING:
Plan to Share IPD: No